CLINICAL TRIAL: NCT06285461
Title: Understanding the Role of Food Intake and Endocrine Factors in Brown Adipose Tissue Function
Brief Title: Food Intake, Endocrine Factors and Brown Fat
Acronym: FoodBAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Kirsi Virtanen, Professor, Turku University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: T2566/2023
Record Dates: First submitted 2024-02-15; First posted 2024-02-29 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Obesity
Keywords: Brown adipose tissue; Gut peptides; Meal-induced thermogenesis; Gut-BAT-brain axis
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This will be a crossover study in which participants undergo two postprandial test days with meals with high- or low-hedonic reward and two weeks of washout between interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-palatable meal (Experimental): Acute intake of a non-palatable meal, i.e., with low-hedonic reward, followed by PET/CT scans with three different radiotracers ([15O]H2O, [15O] oxygen, and [11C]-carfentanil.
  Interventions: Behavioral: Non-palatable meal
- Palatable (Experimental): Acute intake of a palatable meal, i.e., with high-hedonic reward, followed by PET/CT scans with three different radiotracers ([15O]H2O, [15O] oxygen, and [11C]-carfentanil.
  Interventions: Behavioral: Palatable meal

INTERVENTIONS:
Behavioral: Non-palatable meal — Participants will consume a meal that corresponds to 40% of their daily resting metabolic rate and balanced diet but with low hedonic reward.
  Other Names: low-hedonic reward
  Arms: Non-palatable meal
Behavioral: Palatable meal — Participants will consume a meal that corresponds to 40% of their daily resting metabolic rate and balanced diet but with high-hedonic reward.
  Other Names: high-hedonic reward
  Arms: Palatable

SUMMARY:
This study will investigate how the acute intake of foods with high and low hedonic reward differentially affects brown adipose tissue and the interplay between gut peptides, brown fat, and the brain (gut-BAT-brain axis).

DETAILED DESCRIPTION:
Background: The prevalence of obesity is alarmingly high and contributes to the dysfunction of other metabolic organs and tissues, increasing the risk of cardiometabolic diseases. Food products rich in sugar, sodium, and saturated fatty acids, i.e., with high hedonic reward, are shown to disrupt energy homeostasis by overriding the homeostatic control of food intake, promoting body weight gain. Contrary to white adipose tissue, brown adipose tissue uses glucose and triglycerides as fuel to dissipate energy as heat and has been considered an essential target for combating obesity. Recently, it has been shown that meal-induced thermogenesis (MIT) is associated with BAT function and that the postprandial secretion of secretin plays a role in BAT activation and satiety. Therefore, we hypothesize that foods with different degrees of hedonic reward (i.e high-palatable foods) affect the gut-BAT-brain axis, modulating energy homeostasis. Moreover, it differentially affects lean and obese individuals. Methods: This crossover clinical trial consists of two acute postprandial tests (low versus high-hedonic reward meals) with two weeks of washout. Thirty participants (15 lean and 15 with overweight/obesity) will undergo PET/CT scans with short-living radiotracers ([15O]-O2, [15O]-H2O PET/CT) before and after consumption of the two test meals to analyze BAT function. After food intake, one [11C]-carfentanil PET/CT will be carried out to understand the role of the brain in the gut-brain-BAT axis. Before and after the test meal, energy expenditure (indirect calorimetry) and circulating gut peptides will be analyzed to investigate the interplay between gut and BAT. The effect of organoleptic cues on the gut peptides and BAT will also be examined. Participants will answer dietary, behavioral, and physical activity questionnaires at the start of their participation.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females

  * Between 18 and 45 years old.
  * For the lean group: BMI<25.0 kg/m2
  * For the group with overweight/obesity: BMI>27.5 kg/m2 and a waist circumference of over 94 cm (men) or 80 cm (women).

Exclusion Criteria:

* • Inability to have PET/CT (claustrophobia, weight > 150 kg);

  * Pregnancy and pregnancy-related conditions (postpartum/lactation during the last 12 months, or planning to become pregnant soon);
  * Major alterations in the menstrual cycle (e.g., amenorrhea);
  * Use of nicotine-based products;
  * Hypo- or hyper- thyroidism (medical history, TSH, T3 or T4 levels out of the normal range);
  * Diabetes mellitus (fasting Hb1Ac >6.5% or fasting glycaemia>125 mg/dL) or abnormal oral glucose tolerance test (2h OGTT > 7.8 mmol/L);
  * Hypertension (blood pressure > 160/100 mmHg) or abnormal cardiovascular status (arrhythmia and/or long QTc in ECG, abnormal cardiac murmur, previous history of cardiovascular disease);
  * Abnormal coagulopathy (e.g., clotting abnormality);
  * Malignancies, immunological, autoimmune and primary/secondary immunodeficiency disorders (including or not any active treatment).
  * Virus or bacterial infection (both asymptomatic and symptomatic picture) within the 30 days prior to the study start;
  * Episode of fever or major surgery, burns and traumas within the month prior to the study start
  * Chronic infections requiring chronic antibiotic or anti-viral treatment
  * Whole blood donation in the last 3 months (>400 mL of blood) or plans for blood donation during the entire protocol period
  * Weight change (intentional or not) over the last 6-months > than 5% of body weight, or plan to lose weight during the study,
  * Use of any medication that, in the opinion of local clinician/researcher, would negatively affect or mitigate full participation and completion, or could influence the study results. This especially applies to the use of β or α adrenergic receptors agonists/antagonists (e.g., β-blockers). In addition, participants in use of medication for glucose control or weight loss such as GLP-1 analogs will not be included.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Brown adipose tissue metabolism | Fasting and postprandial (30 minutes after the consumption of two different meals, 2 weeks of washout between them)
  Brown adipose tissue metabolism will be assessed using 15O-O2 and 15O-H2O PET/CT, at room temperature, at fasting, after food cues, and after food intake.
Changes in gut peptides | Fasting and postprandial (30, 60, 90, and 120 minutes after meal intake)
  Changes in gut peptides (secretin, GIP, GLP-1) from fasting to postprandial state (after intake of meals with high- or low-hedonic reward).
Differences in μ-opioid receptors in the human brain | The 11C-carfentanil binding potential (BP) will be analyzed 45 minutes after the consumption of the two meals (high or low-hedonic reward). The comparisons will be between the two meals.
  Differences in the brain's μ-opioid receptor (MOR) system (11C-carfentanil binding potential - BP). The differences between the two meals on 11C-carfentanil BP will be analyzed.

SECONDARY OUTCOMES:
Energy expenditure/Meal-induced thermogenesis | Changes in energy expenditure after food intake (30 minutes, 1 hour 30 minutes and 2 hours 30 minutes after food intake)
  Changes in energy expenditure (from indirect calorimetry) after the intake of the two meals will be compared.
Visual Analogue scale (VAS) | Fasting, 30, 60, 90, and 120 minutes after food intake
  Changes in VAS after food intake compared to fasting

CONTACTS AND LOCATIONS:
Overall Officials: Milena Monfort-Pires, PhD, Study Director — University of Turku; Kirsi A Virtanen, Professor, Principal Investigator — University of Turku
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No